CLINICAL TRIAL: NCT05734248
Title: Fractional Laser Drug Delivery of a Local Anesthetic to Mitigate Pain From Filler Injection
Brief Title: Fractional Laser Drug Delivery of a Local Anesthetic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ioannina (Other)
Responsible Party: Principal Investigator, Konstantinos Seretis, Ass. Professor of Plastic Surgery, University Hospital, Ioannina
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Other
Other Study IDs: 00000010
Record Dates: First submitted 2023-02-06; First posted 2023-02-17 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Aging; Face; Atrophy
MeSH Terms: conditions — Facies; Atrophy | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Split-face model
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This test region (right or left cheek) will be pretreated with a fractional carbon dioxide laser (ablative fractional laser; AFL) with a 100 μm spot at 5% density and a pulse energy of 2.5 mJ/microbeam, single pulse at t0 in a operator- and subject- blinded fashion. A lidocaine and tetracaine mixture cream will be applied at each cheek at t1.Ten minutes after cream application (incubation time), the facial filler injections will be performed.
  Interventions: AFL Device: AFL Drug: anesthetic mixture cream
  Interventions: Procedure: Facial filler injection
- Control (Placebo Comparator): A pass with the same fractional carbon dioxide laser with a 100 μm spot at 5% density and a pulse energy of 2.5 mJ/microbeam, single pulse will be given at the area right adjacent to the test region on the other to the intervention cheek ("sham AFL") at t0 in a operator- and subject-blinded fashion.
  A lidocaine and tetracaine mixture cream will be applied at each cheek at t1.Ten minutes after cream application (incubation time), the facial filler injections will be performed.
  Interventions: sham AFL Device: sham AFL Drug: anesthetic mixture cream
  Interventions: Procedure: Facial filler injection

INTERVENTIONS:
Procedure: Facial filler injection — Hyaluronic acid will be injected on the cheek, based on the aesthetic evaluation of the face.
  Other Names: hyaluronic acid injection

SUMMARY:
The purpose of this study is to assess the clinical efficacy of fractional CO2 laser-assisted delivery of a topically applied anesthetic to the perceived pain during filler injection.

DETAILED DESCRIPTION:
Rationale: In daily practice, common aesthetic and laser procedures of the face are carried out under local anesthesia using topical formulations. This procedure is time-consuming, as the anesthetic has to be applied at least one hour before treatment, and is often only partially effective, especially on the face due to increased pain perception. The other option, of infiltration of an anesthetic solution, though effective, is often associated with discomfort, and is not favored during facial procedures (due to changes of the facial landmarks), while it is not tolerated by patients who have needle phobia. In the past years, enhanced and accelerated penetration of various topically applied substances, including photosensitizers, has been proven by pretreatment of the skin with a fractional laser, creating a pattern of microscopic ablation craters. There is also evidence that transdermal anesthetic cream absorption can be increased by fractional laser pretreatment. These outcomes might suggest that adequate local anesthesia may be achieved by applying an anesthetic drug topically on a skin surface pretreated with a fractional laser. However, little is known about the role and efficacy of the fractional laser on topical anesthetic delivery in the clinical setting of facial fillers injection.

Objective: The primary objective of this study is to assess the analgesic effect of fractional carbon dioxide laser-assisted delivery of a topical anesthetic cream (mixture of lidocaine and tetracaine) compared to the application of this anesthetic without fractional laser pretreatment.

Study design: Prospective, double-blinded, randomized, controlled, within subject, study.

Study population: 21 healthy volunteers ≥18 years, who give written informed consent Intervention: In each subject, each cheek region of the subject will be randomly allocated to (1) ablative fractional laser (AFL) pretreatment (5% density, 2.5 mJ/microbeam) followed by topical application of local anesthetic or (2) sham AFL followed by application of local anesthetic. Sham AFL will be done by delivering an AFL pass at the same 5% density and 2.5 mJ/microbeam right adjacent to the region of local anesthetic application on the cheek. After ten minutes incubation time, the typical filler injections procedure will be performed, through the same always entry points.

Subjects will be asked to indicate pain on a visual analogue scale (VAS) from 0-10 (0: no pain; 10: worst imaginable pain) directly after treatment completion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patient is willing and able to give written informed consent
* Patient asks for facial filler injections (hyaluronic acid) to improve the facial aesthetic/ aging signs

Exclusion Criteria:

* History of keloid or hypertrophic scar formation or complicated wound healing
* Presence of any active skin disease
* Known allergy to local anesthesia
* Pregnancy or lactation
* Incompetency to understand what the procedure involves
* Current complaints of chronic pain or other alterations in pain sensation (e.g. due to diabetes mellitus or lepra)
* Current treatment with systemic analgesics or other medication that can influence pain sensation
* Current treatment with anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Pain-Anesthetic effect of AFL | immediately after the intervention/procedure
  Pain evaluation of the injected filler, with a VAS (0 to 10)

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Plastic Surgery Department, Ioannina
  - Swan Clinic, Ioannina

IPD SHARING:
Plan to Share IPD: Undecided